CLINICAL TRIAL: NCT05884255
Title: Randomized, Open, Positive Control Phase III Clinical Trial of Lutetium (177Lu) Oxodotreotide Injection Combined With Standard-dose Long-acting Octreotide Versus High-dose Long-acting Octreotide in the Treatment of Somatostatin Receptor-positive Advanced Gastrointestinal Pancreatic Neuroendocrine Tumors.
Brief Title: An Open-label Phase 3 Study of Lutetium (177Lu) Oxodotreotide Injection in Subjects With Advanced Gastrointestinal Pancreatic Neuroendocrine Tumors.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRFS-Q-2011-301
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-05

CONDITIONS: Advanced Gastroenteropancreatic Neuroendocrine Tumor
MeSH Terms: interventions — Lutetium; Lutetium-177

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: Lutetium (177Lu) Oxodotreotide Injection；long-acting Octreotide
- Treatment group B (Active Comparator)
  Interventions: Drug: long-acting Octreotide.

INTERVENTIONS:
Drug: Lutetium (177Lu) Oxodotreotide Injection；long-acting Octreotide — Lutetium (177Lu) Oxodotreotide Injection combined with standard-dose long-acting Octreotide
  Arms: Treatment group A
Drug: long-acting Octreotide. — High-dose long-acting Octreotide.
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of Lutetium (177Lu) Oxodotreotide Injection in Subjects With advanced gastrointestinal pancreatic neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. 18~75 years old,male or female；
3. ECOG performance status 0 or 1
4. Unresectable locally advanced or metastatic gastrointestinal neuroendocrine tumors ( GEP-NETs ) of low and medium grade ( G1 or G2 ) confirmed by histopathology ;

Exclusion Criteria:

1. Central nervous system metastasis is known. Patients who have previously received treatment ( radiotherapy or surgery ) for brain metastases and have no clinical symptoms can be enrolled if the pre-randomized pre-imaging is confirmed to be stable for at least 24 weeks.
2. There are clinical symptoms or diseases of the heart that are not well controlled.
3. Diabetes ( fasting blood glucose > 2 × ULN ) that cannot be well controlled after optimal medical support treatment.
4. Severe urinary incontinence, hydronephrosis, severe micturition dysfunction or indwelling catheter for any reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by BICR | up to 1 years follow-up

SECONDARY OUTCOMES:
Overall Survival(OS) | up to 5 years follow-up
Objective Response Rate(ORR) | up to 1 years follow-up
Duration of Overall Response(DoR) | up to 1 years follow-up
Disease Control Rate | up to 1 years follow-up
Incidence and severity of AE and SAE | up to 5 years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided